CLINICAL TRIAL: NCT05744011
Title: Effects of Tango on Older People With Dementia. Randomized Controlled Study.
Brief Title: Tango for Older People With Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Burgundy (Other)
Responsible Party: Principal Investigator, France Mourey, Professor, University of Burgundy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CERUBFC-2022-09-29-031
Record Dates: First submitted 2023-02-08; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Old Age; Dementia
Keywords: older adults; cognitive impairment; dance movement therapy; physical performance; tango-therapy; quality of life; well-being; gait
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tango group (Experimental): Tango intervention 2 times/week
  1 hour During 3 months Conducted by care staff who previously received training in therapeutic tango from the University of Burgundy.
  Interventions: Other: Tango intervention
- Physical activity group (Active Comparator): Physical activity intervention 2 times/week
  1 hour During 3 months No music Conducted by physical activity professor assisted by care staff
  Interventions: Other: Adapted Physical Activity

INTERVENTIONS:
Other: Tango intervention — The interventions will be implemented by ABB Reportages and will be carried out by nursing staff who had previously received training in therapeutic tango at the University of Burgundy.
  A dance movement therapist and a musician will accompany the interventions twice a month.
  Participants will attend a 1-hour tango session, twice a week for twelve weeks.
  Other Names: dance-movement-therapy
  Arms: Tango group
Other: Adapted Physical Activity — The intervention will be carried out by an Adapted Physical Activity professor and by nursing staff.
  Music is prohibited during the sessions. Participants will attend a 1-hour APA, twice a week for twelve weeks.
  Other Names: APA
  Arms: Physical activity group

SUMMARY:
Cognitive impairment (CI) is the leading cause of loss of autonomy and has a huge impact on physical performance and quality of life (QOL) in older people. Pharmacological treatments currently available have modest efficacy at best. Dance as both artistic and physical activity, combining emotions, social interaction, and sensory stimulation, therefore appears as a non-pharmacological intervention, which could contribute to the prevention of functional decline.

Among all the existing dances, tango occupies a special place because of the cultural and emotional resonance it carries, but also because of what it leads to motor mobilization (variations in the rhythm of walking, rotation of the belts, weight transfers…). These characteristics seem to make the tango an excellent tool for the rehabilitation of balance and gait, as well as for the prevention of the loss of autonomy in older adults with CI.

The objective of this study is to evaluate and compare the effectiveness of an intervention based on tango and classical physical activity.

DETAILED DESCRIPTION:
CI is a major cause of loss of independence in older people. Alterations in balance and gait are very often present, these worsen the overall condition of the patient and are a sign of poor prognosis. Consequently, the quality of life of the patient and his family is severely affected. The pharmacological treatments currently available aim to alleviate the symptoms. Current data support the modest efficacy of these treatments at best. Non-pharmacological interventions (NPI) are key tools for improving physical performance, functional abilities, cognitive, psychological and social functioning. The benefits of NPIs are observed daily in the field. To be better known, recognized and deployed more widely, it is essential to evaluate their effects and their implementation in a scientific way by following the criteria of evidence-based medicine. Dancing is widely appreciated by older people. "It is both an artistic and physical activity that combines emotions, social interaction, sensory stimulation, thus creating enriched environmental conditions for the elderly". Tango in particular has been used as a therapeutic instrument for a long time. Its regular practice has benefits in many aspects of health and can have a positive impact on cognitive abilities, as it requires sustained attention. Studies on tango as a therapy in Parkinson's disease have shown its effectiveness in improving psychomotor and cognitive signs and especially in the quality of life. Numerous studies have demonstrated the benefits that dance-based interventions can bring, far outweighing the risk of falls they represent. From a motor point of view, tango is a moderate-intensity exercise in which static and dynamic postural control is stimulated. This dance, based on walking, proves to be an excellent tool for rehabilitation, prevention of falls, as well as for the prevention of functional decline in older people with CI.

Objectives: The general goal of this project is to analyze the effects of tango on physical abilities, gait and quality of life of older people with C

Secondary objectives:

* Evaluate the effectiveness of this type of program compared to traditional treatment.
* Refine the characteristics of effective management, concerning the dose, frequency, and duration of intervention.
* Analyze the effects of tango on the spatiotemporal parameters of walking.

General hypotheses: Various studies have highlighted the positive effects of tango face of different conditions, including Parkinson's disease. Based on these findings, the investigators hypothesize that tango interventions have a positive effect on physical abilities and quality of life in older adults with CI.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years old
* MMSE < 21
* agreed to participate
* lived permanently in the nursing home
* able to walk 10 meters without human assistance

Exclusion Criteria:

* medical contraindications,
* limited life expectancy
* bedridden persons.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-16 (Estimated); Study Completion 2023-09-29 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline physical abilities (balance, gait speed and lower limbs strength) at 1 and 3 months | Before intervention/ after 1 month / after 3 months
  Physical abilities will be measured with the Short Physical Performance Battery (SPPB). This test is composed of three evaluation criteria: balance, walking speed and sit to stand [23]. Specifically, during the balance test, the subject had to maintain each of three distinct positions for 10 seconds (feet together, semi-tandem and tandem). The failure of a step was the condition to start the second test, in which the subject walked 4 meters two consecutive times. The best score was retained. Finally, the time taken to complete the fastest 5 chair lifts without the help of the upper limbs was evaluated. At the end of the three tests, a score of a maximum of 12 points could be obtained.
Change from Baseline general physical performance at 1 and 3 months | Before intervention/ after 1 month / after 3 months
  The Timed Up & Go test (TUG) is a general physical performance test used to assess mobility, balance and locomotor performance in elderly people with balance disturbances.
  The individual must stand up from a chair (which should not be leaned up against a wall), walk a distance of 3 meters, turn around, walk back to the chair and sit down - all performed at a comfortable and safe pace. One practice trial is permitted to allow the individual to familiarize him/herself with the task. Timing commences with the verbal instruction "go" and stops when the patient returns to seated position. The individual wears their regular footwear and is permitted to use their walking aid (cane/walker) with its use indicated on the data collection form. No physical assistance is given.

SECONDARY OUTCOMES:
Change from Baseline ability to perform activities of daily living (ADL) at 1 and 3 months | Before intervention/ after 1 month / after 3 months
  Ability to perform ADL will be measured using the Katz Index, consisting of a questionnaire assessing abilities in six activities of daily living (ADL): personal hygiene care, dressing, toilet use, locomotion, continence and eating. For each domain, the answer var-ies between: 1 (complete independence), 0.5 (partial independence) or 0 (absolute depend-ence). In total, an index of zero to six is obtained, where zero indicates the highest degree of dependence.
Change from Baseline questionnaire on Quality of Life (QoL) at 1 and 3 months | Before intervention/ after 1 month / after 3 months
  QoL will be measured with the questionnaire Quality of Life in Alzheimer disease (QoL-AD).This questionnaire is administered directly to the participant, up to a severe stage of the disease, and to the main caregiver. The participant and caregiver ratings were combined into a weighted composite score: (2 × patient score + 1 × caregiver score)/3. Thus, the answers provided by the patient remain preponderant in this model. The QoL-AD comprises 13 items (physical health, energy, mood, living situation, memory, family, marriage, friends, self, ability to carry out daily tasks, ability to do things for fun, money and life as a whole). Response options include 1(poor), 2(fair), 3(good) and 4 (excellent), for a total score of 13-52, with higher scores indicating better QoL.
Change from Baseline neuropsychiatric symptoms at 1 and 3 months | Before intervention/ after 1 month / after 3 months
  neuropsychiatric symptoms will be evaluated using the Neuropsychiatric Inventory-Questionnaire (NPI-Q), which is an informant-based interview that assesses neuropsychiatric symptoms of the participant. NPI consists of 10 (or 12) items that are assayed with questions, subquestions, and ratings of frequency and severity.
Change from Baseline signs and symptoms of major depression at 1 and 3 months | Before intervention/ after 1 month / after 3 months
  Signs and symptoms of major depression will be assessed with the Cornell Scale for Depression in Dementia (CSDD), which is a 19-item clinician-administered instrument that uses information from interviews with both the patient and a nursing staff member, a method suitable for demented patients. The scale has high interrater reliability (kw = 0.67), internal consistency (coefficient alpha: 0.84), and sensitivity. Total Cornell Scale scores correlate (0.83) with depressive subtypes of various intensity classified according to Research Diagnostic Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: France Mourey, Professor, Principal Investigator — Inserm U1093, University of Burgundy
Locations (2):
- France (2):
  - Centre Hospitalier du Mont d'Or, Albigny-sur-Saône
  - Ehpad Du Chg Le Val D'Or, Chasselay

REFERENCES:
- [Derived] Bracco L, Pinto-Carral A, Hillaert L, Mourey F. Tango-therapy vs physical exercise in older people with dementia; a randomized controlled trial. BMC Geriatr. 2023 Oct 24;23(1):693. doi: 10.1186/s12877-023-04342-x. PMID 37875856